CLINICAL TRIAL: NCT07399093
Title: Preoperative Evaluation of IVC Collapsibility Index and Caval Aorta Index for Prediction of Hypotension After Induction of General Anesthesia in Patients Undergoing Craniotomy Surgeries
Brief Title: Preoperative Evaluation of IVC Collapsibility Index and Caval Aorta Index After Induction of General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Verina Fares Zaref Bekheet, Assistant Lecturer of Anesthesia, Intensive Care and Pain Management, Ain Shams University, Cairo, Egypt, Ain Shams University
Other Study IDs: FMASU MD08/2024
Record Dates: First submitted 2025-07-24; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Inferior Vena Cava; Collapsibility Index; Caval Aorta Index; Induction; General Anesthesia; Craniotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients scheduled for elective craniotomy surgeries before induction of general anesthesia.
  Interventions: Other: Inferior vena cava collapsibility index; Other: Caval Aorta Index

INTERVENTIONS:
Other: Inferior vena cava collapsibility index — Inferior vena cava (IVC) collapsibility index (IVCCI) will be measured.
  The IVCCI is calculated using the following formula:
  IVCCI = (maximum IVC diameter - minimum IVC diameter) / maximum IVC diameter * 100
Other: Caval Aorta Index — The Inferior vena cava (IVC): Ao index will be derived by taking the ratio of the maximum IVC diameter during expiration and the maximal abdominal aortic diameter during systole.
  - The caval aorta index (IVC/Ao) is calculated using the following formula: IVC/Ao index = IVC diameter / aortic diameter.

SUMMARY:
This study aims to assess the accuracy, repeatability, and reproducibility of preoperative evaluation of Inferior Vena Cava (IVC) collapsibility index and caval aorta index for prediction of hypotension after induction of general anesthesia.

DETAILED DESCRIPTION:
Post- anesthesia hypotension is of common occurrence, and it hampers tissue perfusion. The magnitude of hypotension is determined by the preoperative volume status, which varies depending on American Society of Anesthesiologists (ASA) physical status, preoperative comorbidities, preoperative medications, and fasting.

General anesthesia causes significant alterations in hemodynamics, as both inhalational and intravenous anesthetics cause bradycardia, decrease in systemic vascular resistance and vasodilatation, and decrease in myocardial contractility, cardiac output and stroke volume, with the absence of surgical stimulus, making induction of anesthesia is the most crucial period at which hypotension occurs.

Due to different definitions of hypotension and diverse patient populations, the effect of volume preload on prevention of hypotension is still controversial. Many recommendations to identified sonographic determination of inferior vena cava (IVC) collapsibility index (IVCCI) as non-invasive, and easy technique for evaluating volume status. Recent guidelines from the American Society of Echocardiography support the general use of IVCCI in assessing volume status.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 40 years.
* Both sexes.
* Body Mass Index< 40 kg/m².
* American Society of Anesthesiologists (ASA) physical status I, II.
* Fasted according to the ASA guidelines: 2 hours for clear fluids, 6 hours after light meal, 8 hours after a full meal with high calorie or fat content.
* Scheduled for elective craniotomy surgeries before induction of general anesthesia.

Exclusion Criteria:

* Current or recent pregnancy (within 3 months).
* Pre-existing cardiac disease or hypertension.
* On medications affecting blood pressure [Beta-blockers (BBs) and calcium channel blockers (CCBs)] .
* Refusing to undergo the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This prospective cohort study will be conducted on 40 patients undergoing craniotomy surgeries at Ain Shams University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-01-14 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of ultrasound guided Aorto-Caval index (IVC-AO) | 15 minutes post-induction of general anesthesia.
  Sensitivity of ultrasound guided Aorto-Caval index (IVC-AO) to predict hypotension will be recorded.

SECONDARY OUTCOMES:
Specificity of ultrasound guided Aorto-Caval index (IVC-AO) | 15 minutes post-induction of general anesthesia.
  Specificity of ultrasound guided Aorto-Caval index (IVC-AO) to predict hypotension will be recorded.
Sensitivity of inferior vena cava (IVC) collapsibility index | 15 minutes post-induction of general anesthesia.
  Sensitivity of inferior vena cava (IVC) collapsibility index to predict hypotension will be recorded.
Specificity of inferior vena cava (IVC) collapsibility index | 15 minutes post-induction of general anesthesia.
  Specificity of inferior vena cava (IVC) collapsibility index to predict hypotension will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

DOCUMENTS (1):
  • Study Protocol (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT07399093/Prot_000.pdf